CLINICAL TRIAL: NCT00785759
Title: An Open-label Study to Assess Brain Uptake and Safety of AH110690 (18F) Injection in Subjects With Probable Alzheimer's Disease, Amnestic Mild Cognitive Impairment and Healthy Volunteers
Brief Title: Brain Uptake and Safety With Probable Alzheimer's Disease, Amnestic Mild Cognitive Impairment and Healthy Volunteers
Acronym: ALZ201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry); Medpace, Inc. (Industry); Hvidovre University Hospital (Other)
Responsible Party: Carl G Torres Ph.D., GE Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALZ201
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Alzheimer's Disease; Amnestic Mild Cognitive Impairment
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AH110690 (18F) Injection — All subjects will receive an I.V. dose of [18F]AH110690 (less than 10 mg of total AH110690). The target activity of a single administration of [18F]AH110690 will be 185 MBq (equivalent to a dose of approximately 6 mSv).

SUMMARY:
Study to Assess Brain Uptake and Safety of AH110690 (18F) Injection in Subjects with Probable Alzheimer's Disease, Amnestic Mild Cognitive Impairment and Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* The subject meets National Institute of Neurological and Communicative Disorders and Stroke; Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for clinically probable AD and Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for dementia of Alzheimer's type.
* The subject meets Petersen criteria for amnestic MCI.
* The subject has no evidence of cognitive impairment by medical history.

Exclusion Criteria:

* The subject may not be able to complete the study as judged by the investigator.
* The subject has received ionising radiation exposure from clinical trials in the last 12 months or has participated in any other clinical study within 30 days of study entry.
* The subject has known allergies to [18F]AH110690 or [11C]PIB or their constituents.
* The subject is pregnant or breast-feeding.
* The subject has a history of alcohol and/or drug abuse within the last 2 years based upon a review of medical records.
* The subject has a contraindication for MRI (including, but not limited to, claustrophobia, pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant).
* The subject has a history of head injury with loss of consciousness.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Examine the efficacy and determine visual assessment of raised [18F] brain uptake for separating subjects with probable Alzheimer's Disease from healthy volunteers and assigning amnestic mild cognitive impairment cases to an AD or HV category. | September 2008 - February 2009

SECONDARY OUTCOMES:
Examine the efficacy and parameters of brain [18F] uptake for separating 25 subjects with probable AD from 25 HV, assigning 20 amnestic MCI cases to an AD or HV category by measuring ranges of regional cerebral to cerebellum tracer uptake ratios. | September 2008 - February 2009

CONTACTS AND LOCATIONS:
Overall Officials: Carl G Torres, Ph.D., Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Oslo, Norway